CLINICAL TRIAL: NCT06311604
Title: Evaluation of the Safety of Inhaled Sedation With Isoflurane in Patients With Severe Traumatic Brain Injury
Brief Title: Evaluation of the Safety of Inhaled Sedation With Isoflurane in Head Trauma Patients
Acronym: IsoSAFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC22.0272
Record Dates: First submitted 2023-08-21; First posted 2024-03-15 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Traumatic Brain Injury
Keywords: isoflurane; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Isoflurane

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, single-centre, interventional dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ISOFLURANE SEDATION (Experimental): Inclusions will have 4 phases according to gradual increased doses of isoflurane (0.3 MAC; 0.5 MAC and 0.7 MAC) Upgrading dose of isoflurane in each phase will be validated by an independent data and safety monitoring committee (DSMC).
  Inclusion of 12-15 additional patients will be included at the 0.7 MAC dose, to have 18 patients exposed to 0.7 MAC isoflurane.
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Isoflurane — Inclusions will have 4 phases according to gradual increased doses of isoflurane:
  Phase 1: Inclusion of 3 patients with 0.3 MAC isoflurane. In the absence of an increase of ICP > 20% from baseline, inhaled sedation is maintained for 24 hours until the primary endpoint is assessed. If there one patient who does not tolerate this threshold, three additional patients will be included in this phase. A maximum of one treatment failure (see definition below) is tolerated in the phase 1
  Phase 2: Inclusion of 3 additional patients with isoflurane dosage of 0.5 MAC under the same conditions as phase 1.
  Phase 3: Inclusion of 3 additional patients with isoflurane dosage of 0.7 MAC under the same conditions as phases 1 and 2.
  Phase 4: Inclusion of 12-15 additional patients will be included at the 0.7 MAC dose, to have 18 patients exposed to 0.7 MAC isoflurane.

SUMMARY:
Intensive care management of patient with severe traumatic brain injury (TBI) includes deep and prolonged sedation with intravenous hypnotics (propofol, midazolam, ketamine) in combination with opioids to prevent and/or treat episodes of intracranial hypertension. However, some patients may develop tachyphylaxis with a gradual increase of administered intravenous hypnotics and opioids to maintain the same level of sedation. This situation leads to a failure in controlling intracranial pressure (ICP) and/or to the risk of adverse effects due to high-dose sedatives: haemodynamic instability, prolonged mechanical ventilation, neuromyopathy, delirium, withdrawal syndrome.

Halogenated agents (Isoflurane, Sevoflurane) are a class of hypnotics routinely used in the operating room. However, doses used in surgical patients (> 1 Minimal Alveolar Concentration, MAC) are not suitable in neuro-intensive care unit (ICU) patients at risk of intracranial hypertension because of the cerebral vasodilator effects of halogenated agents at this dosage, hence the risk of high ICP and compromised cerebral perfusion pressure.

The use of halogenated agents has been recently possible in the ICU through dedicated medical devices (Sedaconda ACD, Mirus). Recommended dosage are lower in the ICU, i.e. 0.3-0.7 MAC, because of their association with intravenous hypnotics and the absence of surgical stimuli. Several clinical studies in general ICUs showed improved sedation quality, reduced duration of mechanical ventilation, faster arousal and shorter extubation time, and lower costs in halogenated group compared with control group receiving midazolam or propofol. At low doses, the effects on ICP and intracerebral haemodynamics of halogenated agents are minor according to the available literature. In addition, beneficial effects were found on cerebral ischaemic volume in animal models treated with halogenated agents. However, there is a need to explore the benefit-risk ratio of the use of halogenated agents in the severe TBI population.

The investigator hypothesise that 0.7 MAC Isoflurane can be administered in this population without deleterious effect on ICP.

DETAILED DESCRIPTION:
Intensive care management of patients with severe neurological injury regularly involves deep and prolonged sedation with intravenous hypnotics (propofol, midazolam, ketamine) in combination with morphine, with the aim of preventing and/or treating episodes of intracranial hypertension (ICHT). However, the tachyphylaxis associated with intravenous hypnotics requires a continuous increase in the doses administered to maintain the same level of sedation, or even a combination of several pharmacological classes. This progressive tolerance to hypnotics may result in the failure of the sedation strategy for certain neuro-injured patients and/or expose them to the undesirable effects of high doses of intravenous hypnotics: haemodynamic instability, longer periods of mechanical ventilation, neuromyopathy, mental confusion and withdrawal syndrome.

Inhaled halogens are a class of hypnotics used daily in the operating theatre to maintain anaesthesia. At the doses used in anaesthesia (> 1 MAC - Minimal Alveolar Concentration), they are contraindicated in neuro-injured patients at risk of HTIC because of their cerebral vasodilatory effects, which can lead to an increase in intracranial pressure (ICP) and compromise cerebral perfusion. Halogens (Isoflurane, Sevoflurane) can be used in intensive care with appropriate medical devices (Isoconda, Mirus). They are used at more moderate doses (< 1 MAC) because they are combined with intravenous hypnotics and because there is no surgical stimulus. Several clinical studies in general intensive care have shown improved sedation quality, reduced duration of mechanical ventilation, quicker awakening and shorter time to tracheal extubation, and lower costs in the group treated with a halogenated agent compared with the control group receiving midazolam or propofol. At these low concentrations, the effects on ICP and intracerebral haemodynamics are much less marked, according to the studies published on this subject. In addition, beneficial effects on the volume of cerebral ischaemia have been shown in animal models treated with halogenated agents. However, there is a need for a precise study of the benefit-risk ratio of using halogenated agents in neurological patients.

The Anaesthesia and Intensive Care Unit at the CHUGA has been internationally recognised for many years in the management of sedation-analgesia in intensive care. In connection with this, the experience acquired by the CHUGA's neuro-resuscitation unit in brain monitoring will be used to explore in detail the effects of halogenated agents on intracerebral haemodynamics and intracranial pressure.

the investigator hypothesise that the administration of Isoflurane at 0.7 MAC can be used in this population without deleterious effect on ICP.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Hospitalized in surgical intensive care (CPR and RNC) for severe head trauma
* On intravenous hypnotic therapy for at least 24 hours with at least 2 lines of IV hypnotics and requiring continued sedation for at least 24 hours, with a RASS of between -3 and -5
* Initial ICP < 15 mmHg on introduction of isoflurane
* Functional intracranial pressure sensor
* Transcranial Doppler measurements performed within 24 hours
* Written informed consent from a legal representative/relative/trusted person. In the absence of a legal representative, the patient may be included under the emergency procedure.

Exclusion Criteria:

* Patients who have had a decompressive craniectomy
* Patients with a personal or family history of malignant hyperthermia
* Patients with a history of long QT syndrome
* Patients taking MAOI-type antidepressants (iproniazid (MARSILID) and moclobemide (MOCLAMIDE))
* Patients with known hypersensitivity to isoflurane or other volatile halogenated anaesthetic agents
* Patients who have experienced liver damage, jaundice, unexplained fever, or eosinophilia after administration of a halogenated anaesthetic.
* Patients expected to die within the next 24 hours
* Subject in a period of exclusion from another clinical trial,
* Technical unavailability of the inhaler
* Persons covered by articles L1121-5 to L1121-8 of the CSP (corresponding to all protected persons: pregnant women, women in childbirth, nursing mothers, persons deprived of their liberty by judicial or administrative decision, persons subject to a legal protection measure).
* No European social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of sedation with 0.7 MAC of inhaled isoflurane in cranial trauma patients in terms of intracranial pressure. | 36 hours
  Composite criterion :
  1. Deaths (attributable to isoflurane) at "H+24 target MAC reached".
  2. 2 consecutive hourly averages of ICP > 20 mmHg during the 24 hours after the target MAC has been reached will be considered as a failure.

SECONDARY OUTCOMES:
To assess the effect on cerebral blood flow of inhaled isoflurane sedation in patients with cranial trauma. | 36 hours
  Changes between "before introduction" and "H+24 MAC target reached of transcranial Doppler parameters
To assess the effect on cerebral blood flow of inhaled isoflurane sedation in patients with cranial trauma. | 36 hours
  Changes between "before introduction" and "H+24 MAC target reached of Tissue oxygen pressure if applicable
To assess the effect on cerebral blood flow of inhaled isoflurane sedation in patients with cranial trauma. | 36 hours
  Changes between "before introduction" and "H+24 MAC target reached" in Cerebral Perfusion Pressure = MAP - ICP
To assess the effect on cerebral blood flow of inhaled isoflurane sedation in patients with cranial trauma. | 36 hours
  Changes between "before introduction" and "H+24 MAC target reached" in ICP dose
To assess the extra-neurological effects of inhaled isoflurane sedation in head trauma patients | 36 hours
  Changes between "before introduction", "H+24 target MAC reached" in biology parameters
To assess the extra-neurological effects of inhaled isoflurane sedation in head trauma patients | 36 hours
  Changes between "before introduction", "H+24 target MAC reached" in Dose of noradrenaline; volume of filling fluids administered
To assess the extra-neurological effects of inhaled isoflurane sedation in head trauma patients | 36 hours
  Changes between "before introduction", "H+24 target MAC reached" in DVE: drainage level, drainage volume/24h
To assess the savings in intravenous hypnotics associated with isoflurane inhalation sedation in head trauma patients | 36 hours
  Change between "before introduction" and "H+24 MAC target reached" in the dose of intravenous hypnotics consumed
To assess the feasibility of inhaled sedation with isoflurane in patients with head trauma | 36 hours
  Rate of non-insertion of isoflurane administration device: cause of withdrawal before "H+24 after target MAC reached".
To assess the neurological outcome at D28 after inhaled sedation in head trauma patients | 28 days
  Neurological outcome at D28 assessed using the Glasgow Outcome Scale (GOSe). 1-4 = poor outcome 4-8 = good outcome

CONTACTS AND LOCATIONS:
Overall Officials: barthélémy BERTRAND, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, Choisir Une Région, France

REFERENCES:
- [Background] Meiser A, Volk T, Wallenborn J, Guenther U, Becher T, Bracht H, Schwarzkopf K, Knafelj R, Faltlhauser A, Thal SC, Soukup J, Kellner P, Druner M, Vogelsang H, Bellgardt M, Sackey P; Sedaconda study group. Inhaled isoflurane via the anaesthetic conserving device versus propofol for sedation of invasively ventilated patients in intensive care units in Germany and Slovenia: an open-label, phase 3, randomised controlled, non-inferiority trial. Lancet Respir Med. 2021 Nov;9(11):1231-1240. doi: 10.1016/S2213-2600(21)00323-4. Epub 2021 Aug 26. PMID 34454654
- [Background] Bosel J, Purrucker JC, Nowak F, Renzland J, Schiller P, Perez EB, Poli S, Brunn B, Hacke W, Steiner T. Volatile isoflurane sedation in cerebrovascular intensive care patients using AnaConDa((R)): effects on cerebral oxygenation, circulation, and pressure. Intensive Care Med. 2012 Dec;38(12):1955-64. doi: 10.1007/s00134-012-2708-8. Epub 2012 Oct 25. PMID 23096426
- [Background] Villa F, Iacca C, Molinari AF, Giussani C, Aletti G, Pesenti A, Citerio G. Inhalation versus endovenous sedation in subarachnoid hemorrhage patients: effects on regional cerebral blood flow. Crit Care Med. 2012 Oct;40(10):2797-804. doi: 10.1097/CCM.0b013e31825b8bc6. PMID 22824929
- [Background] Codaccioni JL, Velly LJ, Moubarik C, Bruder NJ, Pisano PS, Guillet BA. Sevoflurane preconditioning against focal cerebral ischemia: inhibition of apoptosis in the face of transient improvement of neurological outcome. Anesthesiology. 2009 Jun;110(6):1271-8. doi: 10.1097/ALN.0b013e3181a1fe68. PMID 19417596
- [Background] Aubanel S, Bruiset F, Chapuis C, Chanques G, Payen JF. Therapeutic options for agitation in the intensive care unit. Anaesth Crit Care Pain Med. 2020 Oct;39(5):639-646. doi: 10.1016/j.accpm.2020.01.009. Epub 2020 Aug 7. PMID 32777434